CLINICAL TRIAL: NCT02276547
Title: Early Feasibility Study of the Neovasc Tiara™ Mitral Transcatheter Heart Valve With the Tiara™ Transapical Delivery System
Brief Title: Early Feasibility Study of the Neovasc Tiara™ Mitral Valve System
Acronym: TIARA-I
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 047-CPT-001
Record Dates: First submitted 2014-10-21; First posted 2014-10-28 (Estimated); Results first posted 2021-05-25 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Mitral Valve Regurgitation
Keywords: Mitral; Regurgitation; Heart valve; Transcatheter; Transapical; Functional; Degenerative; Symptomatic, severe mitral valve regurgitation, high risk for open mitral valve surgery
MeSH Terms: conditions — Mitral Valve Insufficiency; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Transcatheter mitral valve replacement with the TIARA valve and transapical delivery system
  Interventions: Device: Mitral valve replacement

INTERVENTIONS:
Device: Mitral valve replacement — Transcatheter mitral valve replacement
  Other Names: TIARA Mitral Transcatheter Heart Valve, TIARA Transapical Delivery System

SUMMARY:
The purpose of this study is to evaluate the safety and initial performance of the Neovasc Tiara Mitral Transcatheter Heart Valve with the Tiara Transapical Delivery System.

DETAILED DESCRIPTION:
This is an international, multicenter, single arm, prospective, Early Feasibility Clinical Study to evaluate the safety and performance of the Neovasc Tiara Mitral Valve System in subjects with symptomatic severe mitral regurgitation requiring mitral valve replacement who are at high risk for open chest surgery.

A maximum of 30 subjects will be implanted in this study at a maximum of 10 sites. A maximum of 15 subjects will be implanted in the United States.

Subjects satisfying the inclusion criteria and exclusion criteria will be enrolled to receive the Neovasc Tiara Mitral Transcatheter Heart Valve with the Tiara Delivery System via a transcatheter mitral valve replacement (TMVR) procedure.

ELIGIBILITY:
Inclusion Criteria:

* Severe symptomatic mitral regurgitation (Stage D)
* High surgical risk for open mitral valve surgery
* Subject meets the anatomical eligibility criteria for available size(s)
* NYHA Class III or IV heart failure

Exclusion Criteria:

* DMR deemed by the heart team to be operable.
* Prohibitive risk, deemed too frail or listed for cardiac transplant.
* Unsuitable cardiac structure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-12; Primary Completion 2020-01-06 (Actual); Study Completion 2025-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Anson Cheung, MD, Study Chair — University of British Columbia
Locations (10):
- United States (6):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - Henry Ford Health System, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - University of Washington Medical Center, Seattle, Washington
- ZNA Middelheim, Antwerp, Belgium
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Backer O, Piazza N, Banai S, Lutter G, Maisano F, Herrmann HC, Franzen OW, Sondergaard L. Percutaneous transcatheter mitral valve replacement: an overview of devices in preclinical and early clinical evaluation. Circ Cardiovasc Interv. 2014 Jun;7(3):400-9. doi: 10.1161/CIRCINTERVENTIONS.114.001607. No abstract available. PMID 24944303
- [Background] Nishimura RA, Otto CM, Bonow RO, Carabello BA, Erwin JP 3rd, Guyton RA, O'Gara PT, Ruiz CE, Skubas NJ, Sorajja P, Sundt TM 3rd, Thomas JD, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Creager MA, Curtis LH, DeMets D, Guyton RA, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Stevenson WG, Yancy CW; American College of Cardiology; American College of Cardiology/American Heart Association; American Heart Association. 2014 AHA/ACC guideline for the management of patients with valvular heart disease: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Thorac Cardiovasc Surg. 2014 Jul;148(1):e1-e132. doi: 10.1016/j.jtcvs.2014.05.014. Epub 2014 May 9. No abstract available. PMID 24939033
- [Background] Kappetein AP, Head SJ, Genereux P, Piazza N, van Mieghem NM, Blackstone EH, Brott TG, Cohen DJ, Cutlip DE, van Es GA, Hahn RT, Kirtane AJ, Krucoff MW, Kodali S, Mack MJ, Mehran R, Rodes-Cabau J, Vranckx P, Webb JG, Windecker S, Serruys PW, Leon MB; Valve Academic Research Consortium-2. Updated standardized endpoint definitions for transcatheter aortic valve implantation: the Valve Academic Research Consortium-2 consensus document. J Thorac Cardiovasc Surg. 2013 Jan;145(1):6-23. doi: 10.1016/j.jtcvs.2012.09.002. Epub 2012 Oct 16. PMID 23084102
- See also: Company website with product information — http://www.neovasc.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 27
Completed | 23
Not Completed | 4
Not completed — Death | 2
Not completed — Explant | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.6 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  Canada | 18
  Belgium | 5
  United States | 4
NYHA Functional Class [Number; unit: participants] — Class I:Patients with cardiac disease but without resulting limitations of physical activity.Class II:Patients with cardiac disease resulting in slight limitation of physical activity and are comfortable at rest.Class III:Patients with cardiac disease resulting in marked limitation of physical activity and are comfortable at rest.Class IV:Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort.Symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest.If any physical activity is undertaken,discomfort is increased.
  participants
    NYHA Functional Class I | 0
    NYHA Functional Class II | 0
    NYHA Functional Class III | 26
    NYHA Functional Class IV | 1
Predicted Surgical Mortality [Mean (Standard Deviation); unit: Probability Percentage] — The Society of Thoracic Surgeons' risk models predict the risk of operative mortality and morbidity after adult cardiac surgery on the basis of patient demographic and clinical variables. The models are primarily used to adjust for case mix when comparing outcomes across institutions with different patient populations. Such comparisons are provided in the Database reports received by STS Database participants. The STS models are also used by physicians and patients as tools for understanding the possible risks of surgery.
  Probability Percentage | 7.4 (3.7)
Ejection Fraction [Mean (Standard Deviation); unit: Percentage] | 39 (8.3)
Mitral Regurgitation Severity [Count of Participants; unit: Participants] — Measurement assessed by independent echocardiographic core laboratory utilizing quantitative and qualitative assessments. Mitral Regurgitation is graded by None, Trace, Mild, Moderate, Moderate-Severe and Severe.
  Participants
    Severe | 26
    Moderate-Severe | 1
Diabetes [Count of Participants; unit: Participants] | 8
Hypertension [Count of Participants; unit: Participants] | 22
Chronic Lung Disease [Count of Participants; unit: Participants] | 10
Peripheral Vascular Disease [Count of Participants; unit: Participants] | 6
Renal Dysfunction [Count of Participants; unit: Participants] — Population: Data was not collected on 4 treated subjects.
  Participants
    number analyzed (Participants) | 23
    (all) | 14
Obstructive Coronary Artery Disease [Count of Participants; unit: Participants] — Population: Data was not collected on 4 treated subjects
  Participants
    number analyzed (Participants) | 23
    (all) | 18
Previous Coronary Artery Bypass [Count of Participants; unit: Participants] | 9
Previous Percutaneous Coronary Intervention [Count of Participants; unit: Participants] — Population: Data was not collected on 4 treated subjects.
  Participants
    number analyzed (Participants) | 23
    (all) | 11
Previous Valve Replacement or Repair [Count of Participants; unit: Participants] | 7
Heart Failure [Count of Participants; unit: Participants] | 27
Previous Myocardial Infarction [Count of Participants; unit: Participants] | 12
Cardiomyopathy [Count of Participants; unit: Participants] | 16
Previous Clinically Significant Arrhythmia [Count of Participants; unit: Participants] | 23
Prior Pacemaker/ICD/CRT [Count of Participants; unit: Participants] | 15

OUTCOME MEASURES:

1. Primary Outcome: Freedom From All-cause Mortality and Major Adverse Events
Description: Defined as disabling stroke, myocardial infarction, renal failure requiring dialysis, life-threatening bleeding, and cardiac surgical or transcatheter reintervention
Time Frame: From the time of implant procedure to 30 days or hospital discharge (whichever is later)
Population: Analysis population is all participants implanted with the Tiara valve.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 27
Participants | 19

2. Secondary Outcome: Number and Percentage of Subjects With All-cause Mortality, Disabling Stroke, Myocardial Infarction, Renal Failure Requiring Dialysis, Life-threatening Bleeding and Cardiac Surgical or Transcatheter Reintervention
Time Frame: 30 days, 90 days, 180 days and annually to five years
Reporting Status: Not Posted

3. Secondary Outcome: Individual 30 Day Rates of Device and Procedure Related Major Adverse Events
Description: 1. All mortality
  2. All stroke
  3. Residual MR > mild (1+)
  4. Life threatening bleeding
  5. Acute kidney injury Grade 3
  6. New pacemaker/LBBB
  7. Coronary occlusion/myocardial infarction
  8. Urgent/emergent surgery or reintervention
Time Frame: 30 days
Reporting Status: Not Posted

4. Secondary Outcome: Number and Percentage of Subjects With Progression of Heart Failure
Description: Readmission for Heart Failure Need for Heart Failure device implantation Cardiac transplantation Listing for transplantation
Time Frame: One year
Reporting Status: Not Posted

5. Secondary Outcome: Device Success; Delivery and Deployment of the Device in the Correct Position and Retrieval of Delivery Catheter
Description: Mitral regurgitation < moderate (2+) Effective valve orifice area ≥ 1.5 cm2 as assessed by post-procedural echocardiogram Mitral Valve gradient < 5 mmHg No migration No fracture No endocarditis Stroke free No additional valve/access related interventional or surgical procedures
Time Frame: Post procedure, discharge, 30 days, 90 days, 180 days and annually for five years
Reporting Status: Not Posted

6. Secondary Outcome: Performance
Description: Clinical performance as measured by NYHA Functional Class, 6MWT, and the KCCQ Hemodynamic performance as assessed by echocardiography: mean MV gradient, mitral regurgitation, effective orifice area of the MV, LV systolic and diastolic dimensions as well as volume Stroke free survival Original intended device in place No additional valve/access-related interventional or surgical procedures
Time Frame: 30 days, 90 days, 180 days and annually for five years
Reporting Status: Not Posted

7. Secondary Outcome: Days Alive and Out of Hospital
Description: Number of days alive and not hospitalized
Time Frame: At one year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 3/27
Serious Adverse Events (participants affected / at risk) | 19/27
Other Adverse Events (participants affected / at risk) | 6/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=27)
Acute Kidney Injury (Renal and urinary disorders) | 8 (8)
Bleeding (Blood and lymphatic system disorders) | 3 (3)
Stroke/TIA (Nervous system disorders) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 2 (2)
Vascular Access Site and Access Related Complications (Vascular disorders) | 2 (2)
Arrhythmia and Conduction System Disturbances (Cardiac disorders) | 2 (2)
Progression of Heart Failure (Cardiac disorders) | 10 (11)
Decreased Ejection Fraction (Cardiac disorders) | 1 (1)
Infection - Not related to Study Device/Procedure (Infections and infestations) | 5 (6)
Mitral Regurgitation (Cardiac disorders) | 1 (1)
Multi System Organ Failure (General disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Valve Migration (Cardiac disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=27)
Constipation (Gastrointestinal disorders) | 1 (1)
Eye Infection (Eye disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) — No symptoms reported. Troponin increase and ECG changes noted meeting protocol definition. Adjudicated by the CEC as non serious
Pre Syncope (Nervous system disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Adjudicated by the CEC as non serious
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Adjudicated by the CEC as non serious

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT02276547/Prot_SAP_000.pdf